CLINICAL TRIAL: NCT05467137
Title: Sentinel Lymph Node Detection in Patients With Stage Ib-III Melanoma Using MultiSpectral Optoacoustic Tomography (MSOT) and IndoCyanine Green (ICG)
Brief Title: Sentinel Lymph Node Detection in Patients With Stage Ib-III Melanoma Using MSOT and ICG
Acronym: MelanooMSOT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100685
Record Dates: First submitted 2022-07-01; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Melanoma, Stage I; Melanoma, Stage II; Melanoma Stage III
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care + MSOT (Experimental): Standard of care + MSOT
  Interventions: Device: MSOT

INTERVENTIONS:
Device: MSOT — MSOT imaging (after ICG injection)

SUMMARY:
In this study the investigators try to identify the sentinel lymph node in patients with stage Ib-III melanoma in a non-invasive manner without the use of a radioactive tracer by using the new MSOT technology.

DETAILED DESCRIPTION:
Over the past few decades, melanoma has been one of the fastest-growing cancers and the incidence rate of melanoma is still increasing. Standard treatment for melanoma is wide (re)excision. Sentinel lymph node (SLN) biopsy (SLNB) is recommended for patients with melanoma of AJCC stage pT1b or higher according to Dutch guidelines. SLNB provides essential staging information that impacts on the clinical management of patients with melanoma, and the presence of SLN metastasis indicates a significantly worse prognosis. However, the overall complication rate of SLNB is high.

Currently, lymphoscintigraphy using 99mTc-nanocolloid Technetium-99m-nanocolloïd (Tc99m) is the gold standard to identify the sentinel lymph node. However, there are various disadvantages of using 99mTc-nanocolloidTc99m: the involvement of radioisotopes represents a radioactive burden for patients and caregivers, the lymphoscintigraphic imaging has poor spatial resolution, and the involvement of radioisotopes is expensive and creates logistic challenges. Therefore, in this study the goal is to identify the sentinel lymph node in a non-invasive manner without the use of a radioactive tracer. The investigators try to reach this goal by using the fluorophore dye IndoCyanine Green (ICG) and multispectral optoacoustic imaging (MSOT).

MSOT is a new, but increasingly used, imaging modality that has emerged the field of optical imaging. MSOT is based on a highly powerful pulsed laser in different wavelengths. Photo absorbing molecules absorb laser light in a specific wavelength, undergo thermal expansion and create soundwaves which can be detected by special transducers. The MSOT combines conventional ultrasonography with optoacoustic imaging which gives both anatomical and biological information and is currently available in the University Medical Centre Groningen (UMCG).

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade Ib- III melanoma scheduled for SLNB and/or surgical excision.
* Patients must be > 18 years old and be able to give informed consent.
* Skintype I-IV following Fitzpatrick skin classification (MSOT less reliable in skin types >IV)

Exclusion Criteria:

* Apparent hyperthyroidism or autonomous thyroid adenoma of the thyroid gland
* Prior surgery or radiotherapy on involved lymph nodes / area
* Major surgery within 28 days before tracer administration
* Pregnant or nursing women, fertile women will need a negative pregnancy test prior to inclusion
* History of iodine allergy or anaphylactic reactions to insect bites
* Hypersensitivity to ICG or poorly tolerated ICG in the past
* Unexplained allergic reaction in the past
* Skin type >IV following Fitzpatrick skin classification (MSOT less reliable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Concordance rate of SLNs identified by MSOT imaging and ICG versus the standard of care with 99mTc-nanocolloid Tc99m and lymphoscintigraphic imaging | Through study completion (an average of 1 year)

SECONDARY OUTCOMES:
Patient characteristics | Through study completion (an average of 1 year)
  Age, sex, BMI, history and morbidity, localization and extent of primary tumor, baseline blood count/liver and kidney function

CONTACTS AND LOCATIONS:
Overall Officials: van Leeuwen, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided